CLINICAL TRIAL: NCT02149043
Title: Prototype Study on Association Between Clinical, Laboratory and Thermographic Findings in Patients With Ulcerative Colitis
Brief Title: Thermography in Surveillance of Ulcerative Colitis
Acronym: Thermo
Status: Completed | Type: Observational
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Tonći Božin, Gastroenterology Resident, University Hospital Dubrava
Other Study IDs: THERMO-01
Record Dates: First submitted 2014-05-20; First posted 2014-05-29 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Ulcerative Colitis
Keywords: Inflammatory bowel disease; Ulcerative Colitis; Thermography; Endoscopy; CRP; Fecal Calprotectin
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Thermography; Colonoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples for fecal calprotectin concentration measurements.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ulcerative Colitis patients: 30 patients with active ulcerative colitis will be put throe thermography and colonoscopy. Their stool will be tested for fecal calprotectin and their blood for CRP and other laboratory measures.
  Interventions: Device: Thermography; Procedure: Colonoscopy
- Healthy volunteers: 30 healthy individuals matching sex and BMI to those of ulcerative colitis patients will be put throe thermography and have their stool tested for fecal calprotectin and their blood for CRP.
  Interventions: Device: Thermography

INTERVENTIONS:
Device: Thermography — Thermographic imaging of the patient's abdomen surface
Procedure: Colonoscopy — Endoscopic examination of the colon
  Groups: Ulcerative Colitis patients

SUMMARY:
Ulcerative colitis represents a chronic condition occurring in relapsing and remitting fashion with uncertain outcome and requires lifelong treatment with considerable side effects. Diagnostic methods currently in use, clinical (endoscopy), imaging (CT, MR) or laboratory (C - reactive protein, fecal calprotectin) give an insight into disease activity but are possibly associated with significant discomfort for the patient and / or increased risk of irradiation and potential allergic reactions on contrast agents. For that reason there is a need for a noninvasive, biologically inert method for evaluation of disease activity in inflammatory bowel disease (IBD). Thermography possesses most of these characteristics. The aim of this study is to find potential link between pathological thermographic signs and endoscopic findings, serum C reactive protein (CRP) and calprotectin in the stool of patients with active and extensive ulcerative colitis.

DETAILED DESCRIPTION:
Hypothesis: Documenting pathological thermographic signs in patients with extensive ulcerative colitis investigators will demonstrate pathological thermography criteria that correlate with standard inflammatory markers such as Mayo endoscopic subscore (ESS), CRP and calprotectin in patients with ulcerative colitis.

Aims: The aim of this study is to record abdominal thermographic images of patients with active ulcerative colitis (UC), to create interpretational thermographic criteria for these images and to compare them to abdominal infrared (IR) images of healthy volunteers. Furthermore, investigators intend to correlate these criteria with standard markers of inflammation such as CRP and calprotectin in patients with UC at the beginning of treatment and at the end.

Materials and methods: For the purpose of this work, 36 patients with extensive UC and 30 healthy individuals will be put throe thermographic imagining, have their stool tested for calprotectin and their blood for CRP. In addition, patients with UC will receive colonoscopy evaluations.

Expected scientific contribution: The results of this paper would give an additional contribution to existing tools for pursuing ulcerative colitis activity thus demonstrating the potential of thermography as a complementary method to standard methods in assessing disease activity. Establishing diagnostic criteria for this method would be a good addition to present clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopic diagnosis of active extensive ulcerative colitis
* Stool Calprotectin > 150 mcg/g
* CRP > 5 mg/L
* Signed informed consent form

Exclusion Criteria:

* Inability to preform total colonoscopy
* Marked abdominal comorbidities
* Prior abdominal surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited among active ulcerative colitis patients hospitalized in University Hospital Dubrava.
  Healthy individuals matching sex and BMI to those of recruited ulcerative colitis patients.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in abdominal surface temperatures in ulcerative colitis patients at 6 months | Six months
  Patients will be treated with mesalamin, corticosteroids or biologic therapy according to disease status during 6 months. Abdominal temperatures (maximal, minimum and average temperatures measured in Celsius) recorded by a thermographic camera will be acquired at enrollment and after 6 months of therapy.

SECONDARY OUTCOMES:
Correlation of abdominal surface temperatures between ulcerative colitis patients and healthy volunteers. | Baseline and after 6 months
  Comparison of abdominal surface temperatures (maximum, minimum and average) expressed in Celsius between patients with active ulcerative colitis and healthy controls and also between ulcerative colitis patients in remission and healthy controls.
Correlation of abdominal surface temperature values with clinical markers of inflammation in ulcerative colitis. | Baseline and after 6 months
  Maximal, minimal and average abdominal surface temperatures expressed in Celsius will be correlated to the Disease Activity Index (Mayo score). The Index assesses stool frequency (0-3 points, according to severity) rectal bleeding (0-3 points, according to severity), mucosal appearance at endoscopy (0-3 points, according to severity) and physician rating of disease activity (0-3 points, according to severity). All of the points make up a total sum to produce a score ranging from 0 to 12 points (no activity, to most severe activity). All correlations will be performed before and after 6 months of therapy.
Correlation of abdominal surface temperature values with fecal markers of inflammation in ulcerative colitis. | Baseline and after 6 months
  Maximal, minimal and average abdominal surface temperatures expressed in Celsius will be correlated to fecal calprotectin (µg/g) levels. All correlations will be performed before and after 6 months of therapy.
Correlation of abdominal surface temperature values with serum markers of inflammation in ulcerative colitis. | Baseline and after 6 months
  Maximal, minimal and average abdominal surface temperatures expressed in Celsius will be correlated to serum C - reactive protein (mg/L) levels. All correlations will be performed before and after 6 months of therapy.
Correlation of abdominal surface temperature values with endoscopic markers of inflammation in ulcerative colitis. | Baseline and after 6 months
  Maximal, minimal and average abdominal surface temperatures expressed in Celsius will be correlated to endoscopic parameters expressed as Mayo endoscopic subscore on a scale 0 - 3. [0 - normal or inactive disease; 1 - mild disease (erythema, decreased vascular pattern, mild friability); 2 - moderate disease (marked erythema, absent vascular pattern, friability, erosions); 3 - severe disease (spontaneous bleeding, ulceration)].
  All correlations will be performed before and after 6 months of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Marko Banić, MD, PhD, Study Director — University Hospital Dubrava
Locations (1):
- University Hospital Dubrava, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banić M, et al. Thermography in patients with inflammatory bowel disease and colorectal cancer: evidence and review of the method. Periodicum biologorum 113(4): 439-444, 2011.
- [Background] Božin, Tonći, et al.
- [Background] Banić, Marko, et al.
- See also: University Hospital Dubrava — http://www.kbd.hr
- See also: University of Zagreb — http://www.unizg.hr